CLINICAL TRIAL: NCT01256333
Title: Optimization of Arterial Oxygen Transport by Positive End-expiratory Pressure Variation in Acute Respiratory Distress Syndrome
Acronym: OPTIPEP
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-A00942-37; LOC/10-08
Record Dates: First submitted 2010-12-06; First posted 2010-12-08 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Respiratory Distress Syndrome, Adult
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Despite improving in the treatment of acute respiratory distress syndrome (ARDS), this affection keep an elevate rate of death. The strategy of mechanical ventilation is more and more under definite protocol, following large strength randomized studies. Although, it doesn't exist today element allowing to adjust the level of Positive End-Expiratory Pressure (PEEP) with improvement in patient's survival.

The investigators proposed in this study to determinate the level of PEEP adjust to obtain the better arterial oxygen transport (TaO2). The investigators going to conduct a physiologic, observational, none controlled study. All patients hospitalized in intensive care unit of Pontchaillou hospital with ARDS criteria and without specific exclusion criteria will be included. Primary objective is to looking for the optimum level of PEEP for TaO2.

ELIGIBILITY:
Inclusion Criteria:

* patient presenting a Acute Respiratory Distress Syndrone (ARDS) definite by : acute respiratory failure, bilateral alveolo-interstitial infiltrate on chest radiography, absence of increased left ventricular filling pressure, partial pressure of oxygen in arterial blood (PaO2)/Fraction of inspired oxygen(FiO2) <200 and Positive End-Expiratory Pressure (PEEP) > or equal to 5 cmH2O
* Need to invasive mechanical ventilation
* Precedent criteria persisting at least 6 hours
* Haemoglobin > 8g/dl
* Ramsay score at 6

Exclusion Criteria:

* Participation to en other study on the Acute Respiratory Distress Syndrone (ARDS) with the same end-point
* Presence of external circulatory assist
* Left Ventricular Ejection fraction (LVEF)or Left ventricular shortening fraction (LVSF)< 40% after correction of hypovolemia and/or vasoplegia
* Infusion of inotrope
* Presence of Acute Pulmonary Heart
* Following procedure : ExtraCorporeal Membrane Oxygenation(ECMO), prone position, inhalation of Nitrogen dioxyde
* Presence of a chest tube
* Pregnant or nursing mother
* Less than 18 years old
* Complete arrhythmia by atrial fibrillation
* Person under justice protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute respiratory distress syndrome
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-01

PRIMARY OUTCOMES:
Determinate the Positive End-Expiratory Pressure (PEEP) level achieving the best arterial oxygen transport (TaO2) | 1 year

SECONDARY OUTCOMES:
Evolution of pulmonary gas exchanges | 1 year
Evolution of respiratory mechanism parameters | 1 year
evolution of circulatory parameters and needs of catecholamine during the study | 1 year
Appearance of secondary effects due to mechanical ventilation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Loic Chimot, Study Director — CH de Périgueux
Locations (2):
- France (2):
  - Perigueux Hospital, Périgueux, Aquitaine
  - Rennes University Hospital, Rennes, Britanny